CLINICAL TRIAL: NCT02116842
Title: Comparison of the ED95 Dose of 0.075% and 0.1% Bupivacaine for Labour Analgesia in Primigravida.
Brief Title: Minimum Effective Dose (MED) & Epidural Bupivacaine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Collaborators: National Institute of Academic Anaesthesia (NIAA), UK (Unknown); Obstetric Anaesthetists' Association United Kingdom (Other)
Responsible Party: Principal Investigator, Neville Young, Sponsor Quality Assurance Manager, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN10/9307; 2010-020020-21 (EudraCT Number); 11730 (Other: UKCRN)
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Pregnancy; Labour; Primigravida Labour; Epidural Block
MeSH Terms: interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.075% bupivacaine (Experimental): Consenting patients randomised to receive 0.075% bupivacaine and 40 µg fentanyl.
  Interventions: Drug: 0.075% bupivacaine; Drug: 40 µg fentanyl
- 0.1% bupivacaine (Experimental): Consenting patients randomised to receive 0.1% bupivacaine and 40 µg fentanyl.
  Interventions: Drug: 0.1% bupivacaine; Drug: 40 µg fentanyl

INTERVENTIONS:
Drug: 0.1% bupivacaine — Epidural block in early labour.
  Arms: 0.1% bupivacaine
Drug: 0.075% bupivacaine — Epidural block in early labour.
  Arms: 0.075% bupivacaine
Drug: 40 µg fentanyl — Given with different doses of bupivacaine in epidural block.

SUMMARY:
Local anaesthetics are highly toxic drugs. They can cause toxicity by an absolute overdose, accidental injection in a blood vessel or slow absorption from the area of injection. The risk of toxicity when performing regional anaesthesia can be reduced significantly by injecting the optimal dose of local anaesthetic at the correct site.

To date most of the local anaesthetic dose finding studies for epidural labour analgesia has focused on ED50 ( the dose effective in 50% of patients). The purpose of this research study is to find out the ED95 dose (the dose effective in 95% of patients) of local anaesthetic for epidural analgesia in labour.

The dose determined from this research trial will guide the anaesthetists to the optimal starting dose of the local anaesthetics for epidural analgesia in labour. This would lead to decreased chances of toxicity and will improve patient safety.

We aim to recruit a total of 100 pregnant patients in early labour (cervical dilatation ≤ 5 cm) requesting epidural analgesia to answer the research question based on the continual reassessment method. Patients will be recruited according to well-defined criteria. They will be fully informed about the study and have the choice of not participating or opting out at any time during the study. It is not going to affect the kind of treatment they receive. The experts in the field with full safety precautions will perform this study at St James' Hospitals, Leeds.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) 1-3 patients
* Primigravida (1st pregnancy) patients requesting epidural analgesia in early labour (≤ 5 cm cervical dilatation.

Exclusion Criteria:

* Primigravida (1st pregnancy) patients requesting epidural analgesia in late labour (> 5 cm cervical dilatation)
* Multigravida patients ( ≥ 2nd pregnancy)
* ASA > 3
* Allergy to Bupivacaine
* Unable to give written informed consent
* BMI >35
* Abnormal blood coagulation profile
* Patients taking any medication that are indicated in the Summary of Product Characteristics (SPC) as not recommended

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Effective dose in 95% of patients (ED95) dose of bupivacaine for a primigravida in early labour. | up to 30 minutes
  To find out the ED95 dose of bupivacaine 0.075% and 0.1% for epidural analgesia for a primigravida in early labour .

CONTACTS AND LOCATIONS:
Overall Officials: Professor Philip M Hopkins, Principal Investigator — University of Leeds
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom